CLINICAL TRIAL: NCT06299410
Title: An Open-label, Positron Emission Tomography Study to Evaluate Brain Receptor Occupancy, Safety, Tolerability, and Pharmacokinetics After a Single Sublingual Administration of ITI-1284 in Healthy Subjects
Brief Title: PET Study to Evaluate Brain Receptor Occupancy, Safety and Pharmacokinetics of ITI-1284 in Healthy Subjects
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Intra-Cellular Therapies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ITI-1284-008
Record Dates: First submitted 2024-03-01; First posted 2024-03-07 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Intervention Model Description: This study includes up to 3 sequential parts (Parts A, B and C). Within Parts A and B, subjects will be assigned to 1 of 2 cohorts, will receive a single dose of ITI-1284, and undergo one postdose PET/CT scan. In Part C (optional), subjects will receive a single dose of ITI-1284 and undergo up to 3 postdose PET/CT scans.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort A1: 10 mg ITI-1284 (Experimental): Radioligand: [11C]-raclopride
  Interventions: Drug: ITI-1284 10 mg
- Cohort A2: 20 mg ITI-1284 (Experimental): Radioligand: [11C]-raclopride
  Interventions: Drug: ITI-1284 20 mg
- Cohort B1: 20 mg ITI-1284 (Experimental): Radioligand: [11C]-MDL100907
  Interventions: Drug: ITI-1284 20 mg
- Cohort B2: 20 mg ITI-1284 (Experimental): Radioligand: [11C]-DASB
  Interventions: Drug: ITI-1284 20 mg
- Cohort C: 20 mg ITI-1284 (Experimental): Radioligand: [11C]-MDL100907 or [11C]-raclopride
  Interventions: Drug: ITI-1284 20 mg

INTERVENTIONS:
Drug: ITI-1284 10 mg — ITI-1284 tablet
  Arms: Cohort A1: 10 mg ITI-1284
Drug: ITI-1284 20 mg — ITI-1284 tablet
  Arms: Cohort A2: 20 mg ITI-1284; Cohort B1: 20 mg ITI-1284; Cohort B2: 20 mg ITI-1284; Cohort C: 20 mg ITI-1284

SUMMARY:
The study will be conducted as an open-label and single-center study to evaluate the occupancy of ITI-1284 to the dopamine D2 receptor, serotonin 2A (5-HT2A) receptor, and serotonin transporter (SERT) in healthy subjects.

DETAILED DESCRIPTION:
This study consists of up to 3 sequential parts. Part A will evaluate the D2 receptor occupancy for ITI-1284 at two dose levels. Part B will evaluate the 5HT-2A receptor and SERT occupancy for ITI-1284 at one dose level. Part C (optional) will evaluate the time course of receptor occupancy of ITI-1284 on the D2 or 5-HT2A receptor at one dose level.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects between 18 and 50 years old (inclusive);
* BMI inclusive of 18-32 kg/m2 at screening and a minimum weight of 50 kg;
* Willingness to remain in the hospital research unit for the duration of the inpatient period.

Exclusion Criteria:

* Clinically significant abnormality within 2 years of Screening that in the Investigator's opinion may place the subject at risk or interfere with study outcome variables; this includes, but is not limited to, history of or current cardiac, hepatic, renal, neurologic, gastrointestinal, pulmonary, endocrinologic, hematologic, or immunologic disease or history of malignancy;
* Clinically significant abnormal findings in vital sign assessments, supine SBP > 140 mmHg or < 90 mmHg, or supine DBP >90 mmHg or < 50 mmHg or pulse rate > 100 bpm or < 45 bpm at Screening;
* History of psychiatric condition that in the Investigator's opinion may be detrimental to participation in the study;
* Any condition which would preclude MRI or PET/CT examination (eg, implanted metal, claustrophobia, unable to fit in PET/CT or MRI scanners);
* Contraindications based on any previous MRI or the study MRI performed prior to the baseline PET/CT scan.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-04-11 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
% Receptor occupancy | Day 1
  Percent change of binding potential from baseline

SECONDARY OUTCOMES:
Pharmacokinetics: AUC0-t | Day 1
  Area under the plasma drug concentration-time curve (AUC) from time zero to the last measurable concentration
Pharmacokinetics: Cmax | Day 1
  Maximum plasma concentration
Pharmacokinetics: Tmax | Day 1
  Time of maximum plasma concentration
Percentage of subjects with treatment-emergent adverse events | Up to 30 days after the dose of study drug
Change from baseline in ECG QT interval | Day 3
Change from baseline in aspartate aminotransferase | Day 3
Change from baseline in alanine aminotransferase | Day 3

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Site 1, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No